CLINICAL TRIAL: NCT00001123
Title: A Collaborative Double-Blind Placebo-Controlled Trial of Intravenous Ribavirin As a Treatment for Presumed Hantavirus Pulmonary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: 95-066; NCT00004267 (obsolete NCT alias)
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Hantavirus Pulmonary Syndrome
MeSH Terms: conditions — Hantavirus Pulmonary Syndrome | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirin

SUMMARY:
The purpose is to test the safety and effectiveness of intravenous ribavirin therapy in persons with suspected and subsequently proven hantavirus infection. The hantavirus is spread through the air into the lungs when dry rodent feces are moved or disturbed. It is characterized by fever and bleeding.

DETAILED DESCRIPTION:
Patients are randomized to receive either ribavirin or a placebo for 7 days. At the completion of therapy, patients will be seen on follow-up visits on days 14, 28, and 84.

ELIGIBILITY:
Inclusion Criteria:

You may be eligible for this study if you:

* Are 12 years of age or older.
* Are not pregnant.
* Agree to practice sexual abstinence or use accepted barrier methods of birth control/contraception.
* Are not breast-feeding.
* Have a positive blood test for hantavirus.
* Have symptoms suggestive of hantavirus illness.

Exclusion Criteria:

You will not be eligible for this study if you:

* Have severe low blood count (anemia).
* Have a diagnosis of other respiratory viruses (influenza, RSV, etc.).
* Have group A Streptococcus with symptoms of streptococcal pharyngitis, a positive culture from a normally sterile site, or symptoms of bacterial pneumonia.
* Are HIV positive.
* Have cancer.
* Have had any period of irregular heartbeat.
* Have had chemotherapy or other drugs that suppress the immune system within 30 days.
* Have taken by mouth or injection any antiviral drug (other than acyclovir, famciclovir, amantadine or rimantadine.)
* Have taken by mouth or injection corticosteroids equivalent to approximately 0.5 mg/kg prednisone.
* Have taken any experimental drug within 30 days prior to enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- NIAID/DMID/CASG Central Unit, Birmingham, Alabama, United States